CLINICAL TRIAL: NCT04503629
Title: A Phase 2,Double-blinded, Double Dummy, Positive Drug, Parallel, Randomised Controlled Multicenter Trial to Evaluate Efficacy and Safety of Anaprazole in Patients With Duodenal Ulcers.
Brief Title: A Phase 2 Randomised Controlled Trial to Evaluate Efficacy and Safety of Anaprazole in Patients With Duodenal Ulcers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3571-DU-2001
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Duodenal Ulcer，DU
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anaprazole Sodium 20mg QD (Experimental): administered orally once every 30-60 minutes before breakfast for 4 weeks
  Interventions: Drug: Anaprazole Sodium
- Anaprazole Sodium 40mg QD (Experimental): administered orally once every 30-60 minutes before breakfast for 4 weeks
  Interventions: Drug: Anaprazole Sodium
- Rabeprazole sodium 10mg QD (Active Comparator): administered orally once every 30-60 minutes before breakfast for 4 weeks
  Interventions: Drug: Rabeprazole sodium

INTERVENTIONS:
Drug: Anaprazole Sodium — Anaprazole Sodium 20mg
  Arms: Anaprazole Sodium 20mg QD
Drug: Anaprazole Sodium — Anaprazole Sodium 40mg
  Arms: Anaprazole Sodium 40mg QD
Drug: Rabeprazole sodium — Rabeprazole sodium 10mg
  Arms: Rabeprazole sodium 10mg QD

SUMMARY:
A phase 2,double-blinded, double dummy, parallel, positive drug, randomised controlled multicenter trial to evaluate efficacy and safety of 4 weeks treatment of Anaprazole 20mg QD, 40mg QD compared with rabeprazole 10mg QD in patients with duodenal ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male and female
2. Has endoscopic diagnosis of active duodenal ulcer(s) (A1 or A2 stage) within 7 days prior to randomization
3. 1 or 2 ulcers, 3-15 mm in diameter.
4. Signed informed concent form

Exclusion Criteria:

1. Has malignancy ulcer or malignancy ulcer not excluded, compouned ulcer, stress ulcer, esophageal erosion and ulcer, reflux esophagitis, Zollinger-Ellison syndrome.
2. Has esophageal and gastric varices；
3. With severe compliaction, such as pyloric obstruction, bleeding (Forrest I, IIa and IIb) or perforation, and etc；
4. Has other gastrointestinal disease (e.g.gastric ulcer), or has history of inflammatory bowel disease (such as Crohn's disease or ulcerative colitis)；
5. Has undergone surgical resection or partly resection of esophageal, stomach or duodenum；
6. Has used Proton Pump Inhibitors(PPIs) within 5 days prior to randomization, or continuous more than 3 days of use of Proton Pump Inhibitors within 2 weeks prior to randomization；
7. Has been treated with triple or quandruple Helicobacter pylori eradication therapy included PPIs within 28 days prior to randomization；
8. Current use the drugs (such as systemic glucocorticoids, non steroid anti-inflammatory drugs, or anticoagulation drugs) which may induce ulcer or ulceric bleeding or continuous more than 3 days of use the drugs (such as systemic glucocorticoids, non steroid anti-inflammatory drugs, or anticoagulation drugs) within 28 days prior to randomization；
9. Laboratory tests performed in screning stage revealed Alanine aminotransferase (ALT) or aspartate aminotransferase (AST): > 1.5 upper limit of normal (ULN);
10. Laboratory tests performed in screning stage revealed thyroid stimulating hormone (TSH)；
11. Woman in pregnancy or lactation period；
12. Plan for pregancy or not willing to contracept with reliable contraception method during study period and within 90 days after the final time of investigational drug administratio；
13. Have alcohol abuse or drug abuse 1 years prior to screening；
14. Has hypersensitivity or allergy to investigatory drug, comparatory drug or related supplements；
15. Has participated or been participating other clinical trials(non-interventional study is excluded)；
16. Has an uncotroled disease, such as has a history of significant central nervous system (CNS), cardiovascular, pulmonary, hepatic, renal, or mental or psychological disorders with drug treatment that,in the opinion of the investigator, would not be suitable for participating this clinical trial.
17. In the opinion of the investigator, the patients with other situation would not be suitable for participating this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
The endoscopic healing rate of duodenal ulcers at week 4. | Treatment of 4 weeks
  The endoscopic ulcer healing rate is defined as the percentage of patients with endoscopic ulcer healed evaluated by investigators.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fisrst Affiliated Hospital of NanChang University, Nanchang, Jiangxi, China

REFERENCES:
- [Derived] Shu X, Zhu Z, Fu Y, Zhang Z, Wang J, Li X, He S, Fan H, Liu S, Zhang G, Tang J, Huang C, Du Q, Wang X, Xu B, Du Y, Chen Q, Wang B, Chen Y, Duan X, Xie Y, Huo L, Hou X, Lu N. Mucosal Healing Effectiveness and Safety of Anaprazole, a Novel PPI, vs. Rabeprazole in Patients With Duodenal Ulcers: A Randomized Double-Blinded Multicenter Phase II Clinical Trial. Front Med (Lausanne). 2021 Jul 14;8:690995. doi: 10.3389/fmed.2021.690995. eCollection 2021. PMID 34336894